CLINICAL TRIAL: NCT03728283
Title: Tissue Changes Following Connective Tissue Grafting and Two-stage Implant Placement. A Randomised Clinical Trial
Brief Title: Implant Placement in Combination With Connective Tissue Grafting
Acronym: CTG_implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Danae A. Apatzidou, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUTh_5/30-09-2014
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Dental Implant Placement
Keywords: connective tissue graft; implant surgery; two-stage implants; mucosa thickness; crestal bone

STUDY DESIGN:
Intervention Model Description: Prospective, randomised, parallel-group, controlled clinical trial (Altman et al. 2001) with allocation ratio 1:1,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Implant placement (Active Comparator): conventional implant placement following the manufacturer's instructions
  Interventions: Other: Implant placement
- Implant and Connective tissue grafting (Experimental): implant placement in combination with connective tissue grafting
  Interventions: Procedure: implant placement in combination with connective tissue grafting

INTERVENTIONS:
Procedure: implant placement in combination with connective tissue grafting — A connective tissue graft of standardised dimensions was harvested from the palate under local anaesthesia and was stabilised over the implant's neck
  Arms: Implant and Connective tissue grafting
Other: Implant placement — Implants were placed following teh manufacturer's instructions
  Arms: Conventional Implant placement

SUMMARY:
Suitable subjects who were in need of implant placement were randomised between two groups; Group-A (NA=23) received crestal implant placement. In Group-B (NB=23) a CTG harvested from the palate was stabilised over the implant-neck. At the time of implant placement (T0), Groups were categorized as having thin mucosa ≤2.5mm at the surgical site, or thick mucosa >2.5mm. Mucosa thickness, width of keratinised tissue (WKT), crestal bone levels and bone thickness were determined at T0 and at the two-stage surgery (T1).

DETAILED DESCRIPTION:
Initially, 48 patients were recruited from new referrals to the Lab of Preventive Dentistry, Periodontology and Implant Biology, Aristotle University of Thessaloniki (AUTh) for surgical placement of at least one implant located in the upper/lower jaw in the anterior/posterior segment.

Study design An initial screening visit included full-mouth periodontal assessment, radiographic examination, fulfillment of inclusion/exclusion criteria and suitable patients (n=48) were randomised into either treatment Group; in the control Group (Group-A), a conventional surgical protocol was followed for implant placement, while in the test Group (Group-B) implants were placed in conjunction with an autologous CTG. Each Group was further categorized as having thin mucosa (≤2.5mm for Subgroups-AI/-BI) or thick mucosa (>2.5mm for Subgroups-AII/-BII) at the implantation site before implant placement (baseline=T0). Implants were exposed 3-4 months later (T1).

Surgical procedures A single implant system (Osseotite, Certain, parallel wall, Biomet 3i, Florida, USA; implants of 3.25/4.0 mm in diameter) was used in all cases. At T0, following local anaesthesia (lidocaine hydrochloride 2%, epinephrine 1:100000, Lignospan standard, Septodont, France), crestal incisions were performed and full-thickness flaps were raised for implant placement. Implants were placed at the level of the alveolar crest following the manufacturer's surgical guidelines and a two-stage protocol. Flaps were repositioned using absorbable sutures (polygalactic acid 5/0 sutures; PGA, medipac, Greece). In Group-B, a similar protocol was followed as in Group-A, with the exception that following implant placement a CTG was harvested from the palate, between the maxillary canine and the first molar (Liu & Weisgold, 2002) and was stabilised onto the lingual flap using a horizontal mattress suture. Standardised dimensions of the CTG (11×6×1.5mm) were sought to cover the implant's shoulder and extend 3-5 mm on the buccal and the lingual aspect of the alveolar ridge (Fig. 1). Scoring of the periosteum for coronal advancement of the flaps was mainly performed in Group-B (16 of 23 cases).

Post-operative care Post-operative pain and oedema were controlled by Ibuprofen, 600 mg. All participants were prescribed antibiotics (Amoxicillin, 500 mg per 8 hours for 5 days) and were instructed to rinse twice daily with chlorhexidine digluconate (0.12%) and to abstain from oral hygiene in the test area for one week. Any post-operative adverse events (i.e. swelling, suppuration, flap dehiscence, persistent pain) were recorded upon suture removal ten days after surgery.

Clinical assessments

The following clinical assessments were performed at the implant site at T0 and were repeated at T1:

A periodontal probe (Hu-Friedy XP-23/QW) that had an endo-stop attached on it was used to determine the distances which were finally measured in millimetres by a digital calliper (Mitutoyo Europe GmbH) for precision.

Mucosa thickness (mm) was measured by bone sounding on the alveolar crest and at 2- and 4 mm apically, both on the buccal and the lingual aspects.

The WKT (mm) was measured on the mid-buccal aspect of the implant site. The Implant to Bone Crest (I-BC) distance (mm) was measured at four sites, mid-buccally, mid-lingually, mesially and distally and was determined as the distance of the osseous crest from the implant platform.

The Thickness of the buccal and lingual bone (mm) was measured at the level of the implant shoulder and at 3- and 6 mm apically, using a customised metallic calliper (Ustomed, Tuttlingen, Germany). The inner part of one jaw firmly touched the periphery of the screw hole within the implant fixture and the opposing jaw firmly touched the osseous surface of the alveolar ridge at the predetermined depth.

Radiographic assessment Intraoral digital radiography and the VixWin™ Platinum Gendex software (Hatfield, PA, USA) was utilised to linearly assess the I-BC distance on the mesial/distal aspect at T0 and T1. The long-cone paralleling technique was used at a distance of 10 cm between the x-ray head and the digital sensor which was attached to a custom-made silicone bite block for reproducible radiographs.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years of age
* no active periodontal disease (Plaque Index ≤15%, Gingival Index ≤20%, <20% of sites equal to or deeper than 5mm).

Exclusion Criteria:

* medical conditions that contraindicated surgical implant placement,
* medication that interfered with bone metabolism,
* pregnancy or lactation,
* inadequate dimensions of the alveolar ridge or grafted bone at the surgical site,
* tooth extraction 3 months prior to the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Mucosa thickness | implant placement to implant exposure
  measured by bone sounding on the alveolar crest and at 2- and 4 mm apically, both on the buccal and the lingual aspects

SECONDARY OUTCOMES:
Width of keratinised mucosa | Implant placement to implant exposure
  measured on the mid-buccal aspect of the implant site
Implant to Bone Crest (I-BC) distance | Implant placement to implant exposure
  measured at four sites, mid-buccally, mid-lingually, mesially and distally and was determined as the distance of the osseous crest from the implant platform.
Thickness of the buccal and lingual bone | Implant placement to implant exposure
  measured at the level of the implant shoulder and at 3- and 6 mm apically, using a customised metallic calliper (Ustomed, Tuttlingen, Germany). The inner part of one jaw firmly touched the periphery of the screw hole within the implant fixture and the opposing jaw firmly touched the osseous surface of the alveolar ridge at the predetermined depth.
radiographic Implant to Bone Crest (I-BC) distance | Implant placement to implant exposure
  Intraoral digital radiography and the VixWin™ Platinum Gendex software (Hatfield, PA, USA) was utilised to linearly assess the I-BC distance on the mesial/distal aspect at T0 and T1. The long-cone paralleling technique was used at a distance of 10 cm between the x-ray head and the digital sensor which was attached to a custom-made silicone bite block for reproducible radiographs.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Liu CL, Weisgold AS. Connective tissue graft: a classification for incision design from the palatal site and clinical case reports. Int J Periodontics Restorative Dent. 2002 Aug;22(4):373-9. PMID 12212684
- [Derived] Papapetros D, Karagiannis V, Konstantinidis A, Apatzidou DA. Interim tissue changes following connective tissue grafting and two-stage implant placement. A randomized clinical trial. J Clin Periodontol. 2019 Sep;46(9):958-968. doi: 10.1111/jcpe.13159. Epub 2019 Jul 24. PMID 31206749